CLINICAL TRIAL: NCT05487066
Title: Efficacy of ICU-VTE Scale in Predicting Venous Thromboembolism in ICU Patients
Brief Title: Efficacy of ICU-VTE Scale in ICU Patients
Status: Completed | Type: Observational
Sponsor: Lijuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Lijuan Zhang, physician, Wuhan Central Hospital
Organization: Wuhan Central Hospital (Other)
Other Study IDs: WHZXKYL2022-117
Record Dates: First submitted 2022-07-26; First posted 2022-08-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Venous Thromboembolism
Keywords: Venous thromboembolism; Deep vein thrombosis; ICU; Critically ill
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous thromboembolism (VTE) is a common cause of morbidity and mortality among critically ill patients. No uniform standard model of VTE risk for critically ill patients was formatted by now. In 2020, Viarasilpa et al. developed the ICU⁃VTE rating table, mainly for ICU patients. However, it lacks validation. We examined and compared how well the ICU-VTE score predict and stratify VTE risk in comprehensive ICU patients.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a group of thromboembolic diseases including deep vein thrombosis (DVT) and pulmonary thromboembolism (PE), which is a systemic disease caused by a combination of risk factors. The risk of venous thromboembolism can be greatly reduced by the preventive treatment of it in hospitalized patients according to their risk level. The common risk assessment tools for inpatient VTE include the Padua score for medical patients and the Caprini score for surgical patients, but there is no clinical basis for implementing risk assessment for critically ill patients. The question of how to perform VTE risk assessment in ICU patients to prevent and treat the occurrence of VTE is worth exploring.

This study was designed according to a prospective study method. Data and information were collected from the time the patients were admitted to the ICU to the time the patients were discharged from the ICU.There are three purposes for this study. First, to observe the predictive effect and evaluate the value of the ICU-VTE scoring scale in comprehensive ICU patients; Second, to compare the advantages and disadvantages of the ICU-VTE scoring tool with the Padua score (internal medicine) and Caprini score tool (surgery); To analyze the risk factors for VTE in comprehensive ICU patients and to optimize the VTE risk prediction model; Third, to look into the prevention and treatment of VTE in critically ill ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* patients age greater than or equal to 18 years;
* Patients or their family members agreed to the study and signed informed consent.

Exclusion Criteria:

* Patients admitted to ICU with VTE diagnosis or diagnosed with VTE within 24 hours of admission to ICU;
* Use the therapeutic dose of anticoagulation before admission to ICU or within 24 hours in ICU;
* Expected ICU stay of less than 48 hours;
* Patients cannot obtain imaging data to confirm the presence of VTE during ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient in intensive care unit department of Wuhan Central Hospital
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
incidence of VTE | 28-day
  inhospital venous thromboembolism occurrence

SECONDARY OUTCOMES:
all-cause mortality | 28-day
  Death from all causes during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li Zhang, Master, Principal Investigator — Intensive Care Unit, the Central Hospital of Wuhan
Locations (1):
- The Central Hospital of Wuhan, Wuhan, Hubei, China